CLINICAL TRIAL: NCT02575677
Title: Oxycodone in Treatment of Early Labour Pain Efficacy and Safety
Acronym: oksisynnytys
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kuopio University Hospital (Other)
Collaborators: Admescope Ltd (Industry)
Responsible Party: Principal Investigator, Merja Kokki, MD, PhD, Kuopio University Hospital
Other Study IDs: KUH26062012
Record Dates: First submitted 2015-10-08; First posted 2015-10-15 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Labor Pain
Keywords: labor pain; oxycodone
MeSH Terms: conditions — Labor Pain | interventions — Oxycodone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood for the analysis of oxycodone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parturients with oxycodone: Parturients who were given oxycodone
  Interventions: Other: oxycodone

INTERVENTIONS:
Other: oxycodone — oxycodone 0,1/kg up to 10 mg sc.
  Other Names: Ocycodone administration

SUMMARY:
Oxycodone is used to treat early labour pain instead of meperidine. However, the efficacy and effects of oxycodone to the newborn has not been studied. In the present study, patient who has received oxycodone is asked about pain relief and after labour single venous blood sample from the parturient and umbilical cord are taken for the analysis of oxycodone.

ELIGIBILITY:
Inclusion Criteria:

* Oxycodone for pain relief
* age 18 years or more
* given informed consent

Exclusion Criteria:

* no oxycodone
* age less than 18 years
* no informed consent

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parturients who are in early labor and need some pain medication.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2012-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pain measured with numerical rating scale | from the time of oxycodone administration up to the birth of newborn, maximum of 48 hours
  Pain measured with numerical rating scale 0-10 (0=no pain, 10 = worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Merja Kokki, MD, PhD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: No